CLINICAL TRIAL: NCT00938483
Title: A Multicenter, Single-blind, Randomized, Phase II Study of the Tolerability and Safety of NPS-202 in Infants With Clinically Diagnosed Cow's Milk Allergy
Brief Title: Tolerability and Safety of An Infant Formula
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Perrigo Nutritionals (Industry)
Responsible Party: Cynthia Barber, PhD, Vice President, Regulatory, Medical and Clinical Affairs, PBM Products, LLC
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: CTP-0010
Record Dates: First submitted 2009-07-07; First posted 2009-07-14 (Estimated); Last update posted 2009-07-15 (Estimated); Status verified 2009-07

CONDITIONS: Milk Hypersensitivity
Keywords: infant formula; cow's milk allergy
MeSH Terms: conditions — Milk Hypersensitivity | interventions — Infant Formula

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Extensively hydrolyzed infant formula (Experimental): New extensively hydrolyzed formula, NPS-202
  Interventions: Other: Nutramigen Lipil (Infant formula)
- Infant formula - Extensively hydrolyzed Nutramigen Lipil (Active Comparator): Currently marketed extensively hydrolyzed formula (Nutramigen Lipil)
  Interventions: Other: Nutramigen Lipil (Infant formula)

INTERVENTIONS:
Other: Nutramigen Lipil (Infant formula)
  Other Names: Extensively hydrolyed infant formula (Nutramigen Lipil)

SUMMARY:
The purpose of this study is to evaluate an extensively hydrolyzed formula in infants with cow's milk allergy.

ELIGIBILITY:
Inclusion Criteria:

* clinically diagnosed CMA
* </= 12 weeks at time of study entry
* full-term infant
* must be willing to use provided formula as sole source of nutrition
* other than CMA, infant must be otherwise healthy

Exclusion Criteria:

* underlying or confounding gastrointestinal abnormalities
* infants born from an addictive situation, HIV positive
* if parent/guardian is considered likely to be non-compliant with the protocol requirements

Ages: 1 Day to 12 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 108 (Actual)
Dates: Start 2007-08; Primary Completion 2008-09 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Infant reactivity to an extensively hydrolyzed infant formula | 29 days

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia M Barber, PhD, Study Director — Perrigo Nutritionals